CLINICAL TRIAL: NCT04460807
Title: EXemestane in Progesterone and/or Estrogen Receptor Positive Epithelial Ovarian Cancer: A Randomized Phase III Trial, EXPERT
Brief Title: Exemestane in Hormone Receptor Positive High Grade Ovarian Cancer
Acronym: EXPERT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual, COVID 19 emergency and the modification of the standard of care for ovarian cancer treatment
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Federation of Italian Cooperative Oncology Groups (Other)
Responsible Party: Principal Investigator, Andrea DeCensi, Principal Investigator, Ente Ospedaliero Ospedali Galliera
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 56UCS2017; 2018-000693-30 (EudraCT Number)
Record Dates: First submitted 2020-04-27; First posted 2020-07-08 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Ovarian Cancer
Keywords: exemestane; aromatase inhibitors; clinical trial, phase 3; receptors, estrogen; receptors, progesterone
MeSH Terms: conditions — Ovarian Neoplasms | interventions — exemestane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exemestane (Experimental): Standard chemotherapy: paclitaxel 175 mg/m2 + carboplatin AUC 5, on day 1 every 21 days ± bevacizumab 15mg/kg, on day 1 every 21 days. Chemotherapy will be administered for 6 cycles; Bevacizumab will be administered as up to a maximum of 22 cycles. Patients unfit for standard treatment can receive a weekly schedule of treatment or monotherapy with carboplatin alone. Neoadjuvant chemotherapy is allowed in patients unfit for primary elective surgery.
  +
  Exemestane: single oral tablet of 25 mg/day until disease progression, unacceptable toxicity or physician/patient decision to withdraw, whichever comes first.
  Interventions: Drug: Exemestane
- Placebo (Placebo Comparator): Standard chemotherapy : paclitaxel 175 mg/m2 + carboplatin AUC 5, on day 1 every 21 days ± bevacizumab 15mg/kg, on day 1 every 21 days. Chemotherapy will be administered for 6 cycles; Bevacizumab will be administered as up to a maximum of 22 cycles. Patients unfit for standard treatment can receive a weekly schedule of treatment or monotherapy with carboplatin alone. Neoadjuvant chemotherapy is allowed in patients unfit for primary elective surgery.
  +
  Placebo: single oral tablet until disease progression, unacceptable toxicity or physician/patient decision to withdraw, whichever comes first.
  Interventions: Other: Placebo oral tablet

INTERVENTIONS:
Drug: Exemestane — Exemestane in addition to standard therapy, in Experimental arm.
  Other Names: Mestane
  Arms: Exemestane
Other: Placebo oral tablet — Placebo in addition to standard therapy, in Control arm.
  Arms: Placebo

SUMMARY:
In this Italian, multicenter, randomized, double-blind, placebo controlled, phase III study the efficacy of exemestane will be evaluated in addition to the standard front line treatment in patients with hormone-receptor-positive high grade serous or endometrioid Epithelian Ovarian Cancer (EOC). The patients enrolled in the EXPERT trial will receive exemestane or placebo in addition to standard treatment. Patients and investigators will be blinded to study treatment.

The hypothesis underlying the proposed clinical trial is that exemestane added to standard first line therapy will significantly prolong median progression free survival (PFS).

DETAILED DESCRIPTION:
Estrogen and Progesterone play a role in promoting EOC growth, metastasis, and progression. Recent data show that ER and PgR expression is frequent in high grade EOC and has prognostic significance. A large meta-analysis showed a clinical benefit with any endocrine treatment, and in particular for aromatase inhibitors (AIs), with a greatere benefit for ER+ and/or PgR+ patients and platinum sensitive tumors. Moreover, the analysis of a few randomized clinical trials (RCTs) showed a reduced mortality with endocrine therapy in EOC, suggesting that ER and PgR have a predictive role and that inhibition of their activation could therefore be a treatment option for EOC.

Exemestane is a well-tolerated and effective AI in endocrine sensitive breast cancer which inhibits the production of Estrogens by the adipose tissue in postmenopausal women.

In this Italian, multicentre, randomized, double-blind, placebo controlled, phase III study will be assessed the efficacy of exemestane versus placebo in addition to the standard front line treatment in patients with high grade serous or endometrioid EOC, IHC positive (≥ 10%) ER or PgR disease, stage IIB - IV according to the FIGO classification.

The primary objective of the study is to test the superiority of exemestane over placebo in addition to the standard front line treatment in terms of PFS.

Secondary Objectives are:

1. to test whether the percent expression of ER and PgR is predictive of the effect of exemestane on PFS;
2. to test whether the addition of exemestane to the standard front line treatment can prolong Overall Survival (OS);
3. to evaluate objective response rate Overall Response Rate (ORR) of experimental treatment compared with the standard one;
4. to assess whether the effect of exemestane is affected by the proliferative index Ki67;
5. to evaluate the effect of exemestane on Quality of Life (QoL);
6. to evaluate the compliance to the study treatment;
7. to evaluate the safety profile of the experimental treatment compared with the standard one.

Study design: a total of 468 subjects (234 per Arm) will be randomized in a 1:1 ratio to receive either standard chemotherapy treatment plus exemestane (Experimental arm) or standard chemotherapy plus placebo (Control arm). Exemestane/placebo will be self-administered as a single oral tablet of 25 mg/day until disease progression, unacceptable toxicity or physician/patient decision to withdraw, whichever comes first. Radiological disease assessments and CA125 will be performed at baseline and every 4 months from randomization, until end of study or disease progression whichever comes first. Safety assessments will be performed at each cycle during standard chemotherapy treatment, then at each study visit, up to 30 days after the last Experimental Treatment administration.Quality of Life will be assessed by a menopause-specific questionnaire, administered to patients at baseline (T0), at 12 months (T1) and at disease progression (T2). For patients who have signed the specific informed consent, tissues and blood samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Citologically or histologically confirmed high grade serous or endometrial epithelial ovarian cancer, including cancer of fallopian tube and peritoneum. For patients who are candidates for neoadjuvant chemotherapy, diagnosis must be documented via imaging or a core tissue (not fine needle aspiration) biopsy.
* Disease stage IIB to IV according to FIGO classification. For patients who are candidates for neoadjuvant chemotherapy, stage IIB-IV should be documented via imaging or a core tissue (not fine needle aspiration) biopsy.
* Patients must have completed a surgical debulking procedure, or be candidates for neoadjuvant chemotherapy. For patients enrolling after debulking surgery, randomization should occur at a maximum of 12 weeks and not before 4 weeks after surgery.
* Immunoistochemically determined positivity (≥ 10%) for Progesterone and/or Estrogen receptor expression, including determination on cytology smears from ascitic fluid if surgery is differed.
* Measurable or evaluable disease confirmed by radiological imaging, or histological proven ovarian cancer in the absence of postoperatively measurable or evaluable lesions
* Eastern Cooperative Oncology Group - performance status (ECOG-PS) 0-2.
* Written, informed consent obtained prior to any study-specific procedures.

Exclusion Criteria:

* Previous systemic therapy for ovarian cancer.
* Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.
* Inadequate bone marrow, hepatic or renal functions, assessed within 7 days prior to randomization.
* Treatment with hormonal contraceptives during the previous 3 months from diagnosis.
* Concurrent comorbidities, which contraindicates the administration of chemotherapy, or endocrine therapy.
* Pregnant or lactating patients.
* Inability or unwillingness to swallow tablets.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Enrollment: 23 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 20 months
  PFS id defined for each patient as the time from the date of randomization to the date of local or regional relapse, distant metastasis, second primary malignancy or death from any cause, whichever comes first. Patients not recurred, progressed or died while on study or lost to follow-up will be censored at their last disease assessment date.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 20 months
  OS is defined for each patient as the time from the date of randomization to the date of death from any cause. Patients not reported as having died at the end of the study will be censored at the date they were last known to be alive.
Objective Response Rate (ORR) | a CT-scan will be performed every 4 months. Up to 20 months from last patients randomized
  ORR is defined as the number of patients who will experience a complete or partial response divided by the number of patients randomized with at least one target lesion at baseline. Each patient will be assigned the best response ever recorded during the trial
Quality of Life: Menopause Quality of Life (MENQoL) questionnaire | Up to 20 months
  The effect of study treatment will be assessed based on the MENQOL intervention questionnaire based on 29 items divided in four domains (vasomotor, physical, psychosocial and sexual), each scored from 1 to 8 (1 means no symptom, 2 presence of the symptoms but not bothersome, 3-8 an increasing grade of discomfort). Mean changes from the baseline domain scores between treatment arms will be evaluated.
Compliance - Number of administered cycles | Up to 20 months
  Number of administered cycles
Compliance - Reasons for discontinuation and treatment modification | Up to 20 months
  Number of patients for each reasons
Compliance - Dose intensity | Up to 20 months
  Number of tablets taken (i.e., number of tablets given-number of tablets returned)/number of tablets that should have been taken during the treatment period.
Safety (Adverse Events) | Up to 20 months
  Maximum toxicity grade experienced by each patient for each toxicity, proportion of patients experiencing grade 3-4 toxicity for each toxicity, type, frequency and nature of serious adverse events (SAEs).
  * Proportion of patients with at least one SAE.
  * Proportion of patients with at least one serious adverse drug reaction (SADR).

OTHER OUTCOMES:
Circulating and tissue biomarkers | Up to 20 months
  To collect and store blood and tissue samples to create a bio-bank for the assessment of circulating and tissue biomarkers with potentially prognostic/predictive value, including the androgen receptor (AR) expression and the generation of a somatic genomic and transcriptomic atlas of epithelial ovarian cancers, to map the different molecular vulnerabilities lagging behind the single definition of each histological subtype. Data generated will allow to select molecular biomarkers with prognostic/predictive relevance, to have information of patients risk of relapse or to guide novel treatment approaches.
  These biomarker endpoints will be considered in a second phase of the study, if additional funds are available to perform the analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea DeCensi, Principal Investigator — E.O. Ospedali Galliera Genova
Locations (47):
- Italy (47):
  - AO SS Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - Ospedale Oncologico IRCCS Bari, Bari, BA
  - Ospedale degli Infermi, Biella, BI
  - AULSS 1 Dolomiti - Ospedale "Santa Maria del Prato", Feltre, BL
  - Azienda Ospedaliero Universitaria Policlinico S.Orsola-Malpighi, Bologna, BO
  - ASST degli Spedali Civili di Brescia, Brescia, BS
  - Fondazione Poliambulanza, Brescia, BS
  - Ospedale di Manerbio, Manerbio, BS
  - AOU Cagliari, Policlinico Universitario, Cagliari, CA
  - Ospedale Policlinico "SS. Annunziata", Chieti, CH
  - Azienda Sanitaria Locale CN2, Alba, CN
  - Azienda Ospedaliera S.Croce e Carle, Cuneo, CN
  - Ospedale di Mondovì CN1, Mondovì, CN
  - Ospedale Sant Anna di Como, Como, CO
  - ARNAS Garibaldi, Catania, CT
  - Azienda Ospedaliera per l'emergenza Cannizzaro, Catania, CT
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) IRCCS, Meldola, FC
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - ASL 3 Ospedale Villa Scassi, Genova, GE
  - IRCCS AOU San Martino - IST, Genova, GE
  - ASST Lecco - Ospedale "A. Manzoni", Lecco, LC
  - Ospedale "Vito Fazzi", Lecce, LE
  - UOS Oncologia Ginecologica, Ospedale S. Gerardo, Monza, MB
  - Presidio Ospedaliero Unico Av3, Macerata, MC
  - Istituto Europeo di Oncologia (IEO), Milan, MI
  - AOU Policlinico di Modena, Modena, MO
  - A.R.N.A.S. Ospedali Civico Di Cristina Benfratelli, Palermo, PA
  - Ospedale "Guglielmo da Saliceto", Piacenza, PC
  - Azienda Ospedaliero-Universitaria Pisana, Pisa, PI
  - CRO Centro di Riferimento Oncologico, Aviano, PN
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - Azienda Ospedaliera Regionale San Carlo, Potenza, PZ
  - Ospedale "degli Infermi", Faenza, RA
  - Ospedale "Umberto I", Lugo, RA
  - Ospedale Santa Maria delle Croci, Ravenna, RA
  - Azienda Ospedaliera Arcispedale Santa Maria Nuova, Reggio Emilia, RE
  - Policlinico Umberto I, Università di Roma "La Sapienza", Roma, RM
  - Policlinico Universitario Fondazione Agostino Gemelli, Roma, RM
  - ASST Valtellina e Alto Lario, Sondrio, SO
  - Azienda Ospedaliero Universitaria di Sassari, Sassari, SS
  - Fondazione del Piemonte per l'Oncologia - IRCCS, Candiolo, TO
  - AO Ordine Mauriziano, Torino, TO
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza - Ospedale Ostetrico Ginecologico Sant'Anna, Torino, TO
  - Presidio Ospedaliero S. Andrea, Vercelli, VC
  - Medical Oncology Division, Ente Ospedaliero Ospedali Galliera, Genova
  - Istituto Nazionale Tumori - IRCCS "Fondazione G.Pascale", Napoli
  - Azienda Ospedaliero-Universitaria Maggiore della Carità, Novara

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication of the trial will be shared (text, tables, figures, and appendices), after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared 3 months following the publication of the article and they will remain available for 36 months.
Access Criteria: the investigators who would like to use the data have to prepare a proposal that needs to be approved the Steering committee. The aim of the access to study data needs to be specified in the proposal. Proposals should be sent to the Principal investigator (andrea.decensi@galliera.it). To gain access, data requestors will need to sign a data access agreement.